CLINICAL TRIAL: NCT06089642
Title: Virtual Reality Therapy for Pain Management at the Emergency Department
Acronym: VRxOPUS-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114609
Record Dates: First submitted 2023-09-19; First posted 2023-10-18 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-09

CONDITIONS: Pain, Acute
Keywords: Virtual reality therapy; Pain at rest; Emergency department
MeSH Terms: conditions — Acute Pain; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care
- Virtual Reality therapy (Experimental): Patients receive virtual reality therapy in the form of active distraction or focussed attention (randomized between those two)
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — Virtual reality based on distraction and Virtual Reality based on focussed attention
  Arms: Virtual Reality therapy

SUMMARY:
Rationale: Prescriptions of analgesics, especially opioids, have doubled in the Emergency department (ED) over the past decades in response to frequently reported undertreatment of pain in ED patients. Consequently, there is a shift towards a more restrained utilisation of opioids at the ED. However, there are still few (non-)pharmacological alternatives.

Virtual Reality (VR) therapy is a relatively new and promising technique in non-pharmacologic pain reduction and anxiolysis and shows positive results on pain relief and pain.

Objective: Primary objective is to investigate the effect of VR on patient-reported pain outcomes in the ED. Secondary objectives are to investigate the effect of VR on analgesics use, patient-reported outcomes, and process indicators and to identify barriers to implementation. Last, subanalyses will be performed to compare the effectiveness of two types of VR: VR based on distraction (VRD) and VR based on focussed attention (VRF).

Study design: randomized controlled trial.

Study population: Adults admitted to the ED with a NRS pain score of 4 (out of ten) or more and unacceptable pain.

Intervention: There will be a control group receiving usual care and a intervention group that receives additional VR therapy.

Main study parameters/endpoints: The main study outcome is the difference in patient-reported NRS pain score.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥16 years admitted to ED
* NRS pain at rest score ≥4
* Pain not acceptable for patient
* Patient is willing and able to comply with the study protoc

Exclusion Criteria:

* Patients initially treated by another physician than the emergency physician (EP).
* EMV < 14
* History of dementia, seizures
* Severe hearing/visual impairment not corrected
* Headwounds or damaged skin with which comfortable and hygienic use is not possible.
* Presentation to the ED because of chronic pain (≥3 months) exacerbation
* Chronic opioid use (≥3 months)
* Psychiatric disorders interfering with patients' understanding of the study protocol and informed consent

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
NRS-Pain score at rest | throughout study participation, up to 8 hours
  Pain score before and after administration of VR

SECONDARY OUTCOMES:
NRS anxiety scores | Measured every 30 minutes until discharge of patient to maximal 6 hours
  Anxiety score before and after administration of VR
Oral Morphine Equivalent (OME) | throughout study participation, up to 8 hours
  Dose of morphines adminstered to a patient during their stay at the Emergency Department calculated in OME
Administered analgesics at the ED and type | throughout study participation, up to 8 hours
  registered type and total dose of analgesics administered to patient during the time they stayed at the Emergency Department
Administered non-pharmacological analgesia (e.g. casting, reduction of fracture) | throughout study participation, up to 8 hours
  registered type of non-pharmacological analgesia adminstered during patients' stay at Emergency Department
Acceptability of pain at discharge (yes/no) | Assessed at moment of discharge, up to 6 hours after inclusion
  Acceptability of pain at discharge (yes/no)
Patients desire for analgesics upon admittance and at discharge (yes/no) | Asked at moment of admittance and at discharge, up to 6 hours after inclusion
  Patients desire for analgesics upon admittance and at discharge (yes/no)
NRS immersion score | Assessed at moment of discharge, up to 6 hours after inclusion
  Numeric rating score to measure how immersed patients felt in the VR world
Satisfaction with pain management | Assessed at moment of discharge, up to 6 hours after inclusion
  Numeric rating scale to score satisfaction of patients with pain management
Duration ED visit | throughout study participation, up to 8 hours
  duration ED visit in hours
follow-up of patient | Assessed at moment of discharge, up to 6 hours after inclusion
  registered whether patient is admitted to hospital, discharged home or discharged to other facility
Analgesics prescription by emergency physician | throughout study participation, up to 8 hours
  type and dose of analgesics prescribed by emergency physician
Side effect during VR therapy | evaluated every 30 minutes up to max 6 hours
  Open question
Interview one week after ED admission about patient experiences | approximately one week after ED admission
  Interview one week after ED admission about patient experiences exploring barriers and facilitators to implementation

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data is available upon reasonable request
Supporting Information: Study Protocol